CLINICAL TRIAL: NCT06031194
Title: Pharmacogenomics Effects on High-Dose Methotrexate Clearance in Patients With Diffuse Large B-Cell Lymphoma
Status: Completed | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Timothy Voorhees, Principal Investigator, Ohio State University Comprehensive Cancer Center
Other Study IDs: OSU-22305; NCI-2023-03467 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-08-31; First posted 2023-09-11 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Central Nervous System Lymphoma; Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Participants undergo blood sample collection and have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study evaluates pharmacogenomic effects on high-dose methotrexate clearance in patients with diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify SNPs associated with delayed MTX clearance. II. To explore any association between SNPs and increased toxicity.

OUTLINE: This is an observational study.

Participants undergo blood sample collection and have their medical records reviewed on study.

ELIGIBILITY:
Inclusion Criteria:

* * Adult (age ≥ 18 years at diagnosis)

  * Diagnosis of DLBCL or PCNSL
  * Planned to undergo treatment with HDMTX (≥ 3 g/m^2) at the James Cancer Hospital.

Note: patients with CKD are eligible to participate regardless of eGFR provided the treating physician is planning a dose of HDMTX of at least 3 g/ m^2.

* Ability to provide informed consent.

Exclusion Criteria:

* * Patients with a "currently active" second malignancy that, in the opinion of the principal investigator, will interfere with patient participation, or confound data interpretation

  * Pregnancy (positive serum or urine pregnancy test), lactating or breast feeding
  * Prisoners or incarcerated patients
  * Total bilirubin > 5 mg/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with DLBCL or primary CNS lymphoma planned to undergo treatment with HDMTX (≥ 3 g/m^2) at the James Cancer Hospital
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2025-11-05 (Actual); Study Completion 2025-12-23 (Actual)

PRIMARY OUTCOMES:
SNPs (single nucleotide polymorphisms) associated with delayed MTX clearance | Up to 24 weeks
  Determine the SNPs associated with delayed methotrexate clearance

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Voorhees, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu